CLINICAL TRIAL: NCT03034850
Title: Thrombin Generation and Platelet Activation in Cytoreductive Surgery Combined With Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Thrombin Generation and Platelet Activation in CRS/HIPEC
Status: Completed | Type: Observational
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Sven Van Poucke, Medical Doctor, Anesthesiologist, Emergency Physician, Ziekenhuis Oost-Limburg
Other Study IDs: B37120154199
Record Dates: First submitted 2017-01-12; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Mesothelioma; Peritoneum; Pseudomyxoma Peritonei; Peritoneal Carcinomatosis
Keywords: cytoreductive surgery; hyperthermic intraperitoneal peroperative chemotherapy; platelet function; thrombin generation; thromboelastometry
MeSH Terms: conditions — Mesothelioma; Pseudomyxoma Peritonei; Peritoneal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Cisplatin; Doxorubicin; Ifosfamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRS/HIPEC: Patients with a confirmed histological diagnosis of peritoneal disease treated by cytoreductive surgery (CRS) with hyperthermic intraperitoneal peroperative chemotherapy (HIPEC).
  Interventions: Procedure: CRS/HIPEC

INTERVENTIONS:
Procedure: CRS/HIPEC — The generic surgical approach involved peritonectomy procedures and visceral resections called CRS as described by Sugarbaker (1995). Peritoneal disease burden was assessed using the perito- neal cancer index (PCI), which scores 13 intra-abdominal sites on a scale of 0 (no disease) to 3 (lesion size > 5 cm), thus giving a range of possible scores from 0 to 39. The same team performed the surgical procedure of all included patients. Before connection to the patient, the circuit was filled with dextrose 5% (2 L/m2 body surface area) and warmed to 37°C.
  Other Names: oxaliplatinum; 5-fluorouracil; folinic acid; cisplatinum; doxorubicin; ifosfamide

SUMMARY:
Cytoreductive surgery (CRS) with hyperthermic intraperitoneal peroperative chemotherapy (HIPEC), indicated for patients with peritoneal metastases from digestive or gynecological malignancies alike, demonstrates a considerable impact on hemostatic metabolism, both on platelet and on coagulation level. The potential hemostatic interference in CRS and HIPEC is phase dependent. This study demonstrates the combined use of ROTEM (rotational thromboelastometry), PACT (platelet activation test) and CAT (thrombin generation test) assays during CRS and HIPEC with a follow-up of 7 days postoperative.

DETAILED DESCRIPTION:
The purpose of this study was to quantitatively assess the impact of CRS and HIPEC, on various components of hemostasis. Routine laboratory assays such as activated clotting time, activated partial thromboplastin time, prothrombin time, or platelet count might, as demonstrated previously, insufficiently provide specificity and/or sensitivity to assess coagulation and platelet disorders. Therefore, additionally thrombin generation (TG) was analyzed by the calibrated automated thrombogram assay (CAT). Also, platelet function was quantitatively assessed by the PAC-t-UB assay and rotational thromboelastometry (ROTEM) was used to elucidate the contribution of platelets, intrinsic and extrinsic coagulation pathways in peri-operative bleeding. The hypothesis of this study was that the procedure exposed an increased thrombotic risk, resulting in a faster and increased TG and hyper platelet function?

ELIGIBILITY:
Inclusion Criteria:

* a confirmed histological diagnosis of peritoneal disease (e.g., mesothelioma; pseudomyxoma peritonei; colorectal, ovarian, or gastric peritoneal carcinomatosis of colorectal, ovarian, or gastric cancer origin; or abdominal sarcomatosis); and
* age <80 years; and
* a cardiac, renal, hepatic, and bone marrow function compatible with surgery; and
* informed written consent to participate in the study

Exclusion Criteria:(or)

* inherited coagulation abnormalities,
* active systemic infections,
* interstitial lung disease,
* serious cardiac dysrhythmia or condition, New York Heart Association classification of III or IV, congestive cardiac failure, uncontrolled hypertension (diastolic blood pressure constantly >100 mm Hg, systolic blood pressure constantly > 180 mm Hg).
* inadequate bone marrow function at the beginning of the trial, defined as platelet count less than <150 GPT/L or neutrophil granulocyte count less than <1.5 GPT/L.
* inadequate renal function at the beginning of the trial, defined as GFR less than <60 ml/min,
* inadequate liver function at the beginning of the trial, defined as bilirubin >1.5 times ULN (upper limit of normal), active hepatitis B or C infection,
* female patients who are pregnant or breast feeding
* participation in another therapeutic clinical trial.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This prospective observational pilot study, scheduled between April 2015 and July 2016, included 27 patients from the Ziekenhuis Oost-Limburg, Genk, Belgium, after approval by the local medical ethics committee (Eudract/B nr: B371201524199) and written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Blood loss | From surgical incision to 7 days postoperative
  Blood loss and administration of red blood cells, fresh frozen plasma and platelets. Blood loss is quantitatively assessed based on surgical drainage volume measurements, recorded every hour. Once the surgical drains are removed (average 7 days), blood loss is quantified by hemodynamic instability and abrupt, significant decrease of hemoglobin concentration. Blood loss is assessed from the date of CRS/HIPEC surgery until 7 days postoperative or date of death from any cause, whichever came first.

SECONDARY OUTCOMES:
Red blood cell count | From surgical incision to 7 days postoperative
  EDTA-anticoagulated blood was used for cytometric analysis using a whole blood counter Sysmex XE 2100® (Sysmex,Kobe, Japan) to obtain a whole blood count. (million cells/mcL)
White blood cell count | From surgical incision to 7 days postoperative
  EDTA-anticoagulated blood was used for cytometric analysis using a whole blood counter Sysmex XE 2100® (Sysmex,Kobe, Japan) to obtain a whole blood count. (cells/mcL)
Platelet count | From surgical incision to 7 days postoperative
  EDTA-anticoagulated blood was used for cytometric analysis using a whole blood counter Sysmex XE 2100® (Sysmex,Kobe, Japan) to obtain a whole blood count. (platelets/mcL)
Fibrinogen levels | From surgical incision to 7 days postoperative
  Fibrinogen levels were determined with an ACL-9000 (Diamond Diagnostics, Holliston, MA) coagulation analyser. (g/dL)
Prothrombin Time (PT) | From surgical incision to 7 days postoperative
  Prothrombin time was measured using an ACL-9000 coagulation analyser (sec).
Activated Partial Thromboplastin Time (aPTT) | From surgical incision to 7 days postoperative
  Activated Partial Thromboplastin Time was measured using an ACL-9000 coagulation analyser (sec).
Endogenous Thrombin Potential (Thrombin generation assay (CAT)) | From surgical incision to 7 days postoperative
  TG in plasma, measured with the calibrated automated thrombogram (CAT) . Briefly, 80 μl platelet poor plasma (PPP) was mixed with 20 μl of a mixture containing tissue factor (Dade-Behring) at a final concentration of 1 pM and phospholipid vesicles (f.c. 4 μM 20 mol% phosphatidylserine, 60 mol% phosphatidylcholine and 20 mol% phosphatidyl-ethanolamine, Avanti). To calibrator wells, 20 μl of calibrator (α2macroglobulin- thrombin complex) was added instead of TF and PL. After 10 minutes of incubation at 37°C, thrombin generation was initiated by the addition of 20 μl of the thrombin specific substrate, Z- Gly-Gly-Arg-7-amino-4-methylcoumarin (f.c. 416 μM, Bachem) and CaCl2 (f.c. 16.7 mM). Fluorescence was measured with a Fluoroscan Ascent reader (Thermo Labsystems) and data were analyzed with dedicated software (Thrombinoscope, Stago) [20]. Endogenous thrombin potential (ETP) (nM*min)
Lag Time (Thrombin generation assay (CAT)) | From surgical incision to 7 days postoperative
  TG in plasma, measured with the calibrated automated thrombogram (CAT) . Briefly, 80 μl platelet poor plasma (PPP) was mixed with 20 μl of a mixture containing tissue factor (Dade-Behring) at a final concentration of 1 pM and phospholipid vesicles (f.c. 4 μM 20 mol% phosphatidylserine, 60 mol% phosphatidylcholine and 20 mol% phosphatidyl-ethanolamine, Avanti). To calibrator wells, 20 μl of calibrator (α2macroglobulin- thrombin complex) was added instead of TF and PL. After 10 minutes of incubation at 37°C, thrombin generation was initiated by the addition of 20 μl of the thrombin specific substrate, Z- Gly-Gly-Arg-7-amino-4-methylcoumarin (f.c. 416 μM, Bachem) and CaCl2 (f.c. 16.7 mM). Fluorescence was measured with a Fluoroscan Ascent reader (Thermo Labsystems) and data were analyzed with dedicated software (Thrombinoscope, Stago) [20]. lagtime (LT)(min)
Time-to-Thrombin Peak (Thrombin generation assay (CAT)) | From surgical incision to 7 days postoperative
  TG in plasma, measured with the calibrated automated thrombogram (CAT) . Briefly, 80 μl platelet poor plasma (PPP) was mixed with 20 μl of a mixture containing tissue factor (Dade-Behring) at a final concentration of 1 pM and phospholipid vesicles (f.c. 4 μM 20 mol% phosphatidylserine, 60 mol% phosphatidylcholine and 20 mol% phosphatidyl-ethanolamine, Avanti). To calibrator wells, 20 μl of calibrator (α2macroglobulin- thrombin complex) was added instead of TF and PL. After 10 minutes of incubation at 37°C, thrombin generation was initiated by the addition of 20 μl of the thrombin specific substrate, Z- Gly-Gly-Arg-7-amino-4-methylcoumarin (f.c. 416 μM, Bachem) and CaCl2 (f.c. 16.7 mM). Fluorescence was measured with a Fluoroscan Ascent reader (Thermo Labsystems) and data were analyzed with dedicated software (Thrombinoscope, Stago) [20]. Time-to-Thrombin Peak (TTP)(min)
Thrombin Peak (TP) (Thrombin generation assay (CAT)) | From surgical incision to 7 days postoperative
  TG in plasma, measured with the calibrated automated thrombogram (CAT) . Briefly, 80 μl platelet poor plasma (PPP) was mixed with 20 μl of a mixture containing tissue factor (Dade-Behring) at a final concentration of 1 pM and phospholipid vesicles (f.c. 4 μM 20 mol% phosphatidylserine, 60 mol% phosphatidylcholine and 20 mol% phosphatidyl-ethanolamine, Avanti). To calibrator wells, 20 μl of calibrator (α2macroglobulin- thrombin complex) was added instead of TF and PL. After 10 minutes of incubation at 37°C, thrombin generation was initiated by the addition of 20 μl of the thrombin specific substrate, Z- Gly-Gly-Arg-7-amino-4-methylcoumarin (f.c. 416 μM, Bachem) and CaCl2 (f.c. 16.7 mM). Fluorescence was measured with a Fluoroscan Ascent reader (Thermo Labsystems) and data were analyzed with dedicated software (Thrombinoscope, Stago) [20]. Thrombin Peak (TP)(nM)
P-selectin expression (Platelet activation test (PACT)) | From surgical incision to 7 days postoperative
  Platelet activation was quantitatively assessed in un-processed blood by the PACT (Platelet activation test). Addition of specific agonists to whole blood (granule release capacity and in the aggregation potential of platelets). (1) the protease activated receptor (PAR-1) agonist thrombin receptor activator peptide, (2) the glycoprotein VI (GPVI) agonist collagen-related peptide , and (3) the P2Y12 agonist ADP. The reaction mixtures also contain three antibodies directed against GPIb, activated αIIbβ3 and P-selectin. Flow cytometry was used to distinguish between platelets and other cells on forward and sideward scatter pattern and by gating on the CD42b positive cells. Fluorescent intensity in the FITC gate and PE gate was selected to determine activated αIIbβ3 and P-selectin density, respectively, and results are expressed as median fluorescent intensity (MFI). P-selectin expression(MFI, median fluorescent intensity)
αIIbβ3 activation (Platelet activation test (PACT)) | From surgical incision to 7 days postoperative
  Platelet activation was quantitatively assessed in un-processed blood by the PACT (Platelet activation test). Addition of specific agonists to whole blood (granule release capacity and in the aggregation potential of platelets). (1) the protease activated receptor (PAR-1) agonist thrombin receptor activator peptide, (2) the glycoprotein VI (GPVI) agonist collagen-related peptide , and (3) the P2Y12 agonist ADP. The reaction mixtures also contain three antibodies directed against GPIb, activated αIIbβ3 and P-selectin. Flow cytometry was used to distinguish between platelets and other cells on forward and sideward scatter pattern and by gating on the CD42b positive cells. Fluorescent intensity in the FITC gate and PE gate was selected to determine activated αIIbβ3 and P-selectin density, respectively, and results are expressed as median fluorescent intensity (MFI). αIIbβ3 activation (MFI, median fluorescent intensity)
A5 EXTEM (Rotational thromboelastometry (ROTEM)) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: EXTEM (ref.: 503-05, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands), A5: amplitude of clot firmness 5 min after CT (mm)
A5 FIBTEM (Rotational thromboelastometry (ROTEM)) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: FIBTEM (ref.: 503-06, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands), All samples were measured within 1 h after blood collection. A5: amplitude of clot firmness 5 min after CT (mm)
A5 HEPTEM (Rotational thromboelastometry (ROTEM)) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: HEPTEM (ref.: 503-09, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. A5: amplitude of clot firmness 5 min after CT (mm)
A30 EXTEM (Rotational thromboelastometry (ROTEM)) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: EXTEM (ref.: 503-05, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. A30: amplitude of clot firmness 30 min after CT (mm)
A30 FIBTEM (Rotational thromboelastometry (ROTEM)) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: FIBTEM (ref.: 503-06, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. A30: amplitude of clot firmness 30 min after CT (mm)
A30 HEPTEM (Rotational thromboelastometry (ROTEM)) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: HEPTEM (ref.: 503-09, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. A30: amplitude of clot firmness 30 min after CT (mm)
Alpha EXTEM (Rotational thromboelastometry (ROTEM)) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: EXTEM (ref.: 503-05, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. Alpha (the angle between the baseline and a tangent to the clotting curve through the 2 mm point; degree)
Alpha FIBTEM (Rotational thromboelastometry (ROTEM)) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: FIBTEM (ref.: 503-06, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. Alpha (the angle between the baseline and a tangent to the clotting curve through the 2 mm point; degree)
Alpha HEPTEM (Rotational thromboelastometry (ROTEM)) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: HEPTEM (ref.: 503-09, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. Alpha (the angle between the baseline and a tangent to the clotting curve through the 2 mm point; degree)
Coagulation Time CT EXTEM (Rotational thromboelastometry (ROTEM)) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: EXTEM (ref.: 503-05, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. Coagulation Time (CT): test start until a clot firmness amplitude of 2 mm is reached; sec.
Coagulation Time CT FIBTEM (Rotational thromboelastometry (ROTEM)) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: FIBTEM (ref.: 503-06, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands), All samples were measured within 1 h after blood collection. Coagulation Time (CT): test start until a clot firmness amplitude of 2 mm is reached; sec.
Coagulation Time CT HEPTEM (Rotational thromboelastometry (ROTEM)) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: HEPTEM (ref.: 503-09, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. Coagulation Time (CT): test start until a clot firmness amplitude of 2 mm is reached; sec.
Clot Formation Time CFT EXTEM (Rotational thromboelastometry (ROTEM) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: EXTEM (ref.: 503-05, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands), All samples were measured within 1 h after blood collection. CFT: in seconds indicates the time between 2 and 20 mm clot firmness amplitude is achieved (sec)
Clot Formation Time CFT FIBTEM (Rotational thromboelastometry (ROTEM) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: FIBTEM (ref.: 503-06, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. CFT: in seconds indicates the time between 2 and 20 mm clot firmness amplitude is achieved (sec)
Clot Formation Time CFT HEPTEM (Rotational thromboelastometry (ROTEM) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: HEPTEM (ref.: 503-09, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. CFT: in seconds indicates the time between 2 and 20 mm clot firmness amplitude is achieved (sec)
Maximum Lysis (ML) EXTEM Rotational thromboelastometry (ROTEM) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: EXTEM (ref.: 503-05, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. Maximum Lysis (ML; %): maximum lysis during runtime
Maximum Lysis (ML) FIBTEM Rotational thromboelastometry (ROTEM) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: FIBTEM (ref.: 503-06, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). All samples were measured within 1 h after blood collection. Maximum Lysis (ML; %): maximum lysis during runtime
Maximum Lysis (ML) HEPTEM Rotational thromboelastometry (ROTEM) | From surgical incision to 7 days postoperative
  Thrombus formation was measured by ROTEM (Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Standard assays were used according to the manufacturer's recommendations: HEPTEM (ref.: 503-09, Tem International GmbH c/o Dutch Affiliate, Tilburg, The Netherlands). Maximum Lysis (ML; %): maximum lysis during runtime

CONTACTS AND LOCATIONS:
Overall Officials: Sven Van Poucke, MD, Principal Investigator — Ziekenhuis Oost-Limburg

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data will be available 6 months after inclusion of the last patient by contacting the principle investigator (svanpoucke@gmail.com). Once the results of the study are available and published, all data will be part of the publication.

REFERENCES:
- [Background] Sugarbaker PH. Peritonectomy procedures. Ann Surg. 1995 Jan;221(1):29-42. doi: 10.1097/00000658-199501000-00004. PMID 7826158
- [Background] Elias DM, Ouellet JF. Intraperitoneal chemohyperthermia: rationale, technique, indications, and results. Surg Oncol Clin N Am. 2001 Oct;10(4):915-33, xi. PMID 11641098
- [Background] Van der Speeten K, Govaerts K, Stuart OA, Sugarbaker PH. Pharmacokinetics of the perioperative use of cancer chemotherapy in peritoneal surface malignancy patients. Gastroenterol Res Pract. 2012;2012:378064. doi: 10.1155/2012/378064. Epub 2012 Jun 13. PMID 22778722
- [Background] Urano M, Ling CC. Thermal enhancement of melphalan and oxaliplatin cytotoxicity in vitro. Int J Hyperthermia. 2002 Jul-Aug;18(4):307-15. doi: 10.1080/02656730210123534. PMID 12079586
- [Background] Perez-Ruixo C, Valenzuela B, Peris JE, Bretcha-Boix P, Escudero-Ortiz V, Farre-Alegre J, Perez-Ruixo JJ. Population pharmacokinetics of hyperthermic intraperitoneal oxaliplatin in patients with peritoneal carcinomatosis after cytoreductive surgery. Cancer Chemother Pharmacol. 2013 Mar;71(3):693-704. doi: 10.1007/s00280-012-2060-2. Epub 2012 Dec 30. PMID 23274396
- [Background] Schmidt C, Creutzenberg M, Piso P, Hobbhahn J, Bucher M. Peri-operative anaesthetic management of cytoreductive surgery with hyperthermic intraperitoneal chemotherapy. Anaesthesia. 2008 Apr;63(4):389-95. doi: 10.1111/j.1365-2044.2007.05380.x. PMID 18336490
- [Background] Desantis M, Bernard JL, Casanova V, Cegarra-Escolano M, Benizri E, Rahili AM, Benchimol D, Bereder JM. Morbidity, mortality, and oncological outcomes of 401 consecutive cytoreductive procedures with hyperthermic intraperitoneal chemotherapy (HIPEC). Langenbecks Arch Surg. 2015 Jan;400(1):37-48. doi: 10.1007/s00423-014-1253-z. Epub 2014 Oct 16. PMID 25319432
- [Background] Kajdi ME, Beck-Schimmer B, Held U, Kofmehl R, Lehmann K, Ganter MT. Anaesthesia in patients undergoing cytoreductive surgery with hyperthermic intraperitoneal chemotherapy: retrospective analysis of a single centre three-year experience. World J Surg Oncol. 2014 May 1;12:136. doi: 10.1186/1477-7819-12-136. PMID 24886171
- [Background] Bell JC, Rylah BG, Chambers RW, Peet H, Mohamed F, Moran BJ. Perioperative management of patients undergoing cytoreductive surgery combined with heated intraperitoneal chemotherapy for peritoneal surface malignancy: a multi-institutional experience. Ann Surg Oncol. 2012 Dec;19(13):4244-51. doi: 10.1245/s10434-012-2496-y. Epub 2012 Jul 18. PMID 22805865
- [Background] Cooksley TJ, Haji-Michael P. Post-operative critical care management of patients undergoing cytoreductive surgery and heated intraperitoneal chemotherapy (HIPEC). World J Surg Oncol. 2011 Dec 19;9:169. doi: 10.1186/1477-7819-9-169. PMID 22182345
- [Background] Korakianitis O, Daskalou T, Alevizos L, Stamou K, Mavroudis C, Iatrou C, Vogiatzaki T, Eleftheriadis S, Tentes AA. Lack of significant intraoperative coagulopathy in patients undergoing cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (HIPEC) indicates that epidural anaesthesia is a safe option. Int J Hyperthermia. 2015;31(8):857-62. doi: 10.3109/02656736.2015.1075606. Epub 2015 Oct 8. PMID 26446799
- [Background] Falcon Arana L, Fuentes-Garcia D, Roca Calvo MJ, Hernandez-Palazon J, Gil Martinez J, Cascales Campos PA, Acosta Villegas FJ, Parrilla Paricio P. Alterations in hemostasis during cytoreductive surgery and hyperthermic intraperitoneal chemotherapy in patients with peritoneal carcinomatosis. Cir Esp. 2015 Oct;93(8):496-501. doi: 10.1016/j.ciresp.2015.01.012. Epub 2015 Apr 14. English, Spanish. PMID 25882334
- [Background] Kusamura S, Moran BJ, Sugarbaker PH, Levine EA, Elias D, Baratti D, Morris DL, Sardi A, Glehen O, Deraco M; Peritoneal Surface Oncology Group International (PSOGI). Multicentre study of the learning curve and surgical performance of cytoreductive surgery with intraperitoneal chemotherapy for pseudomyxoma peritonei. Br J Surg. 2014 Dec;101(13):1758-65. doi: 10.1002/bjs.9674. Epub 2014 Oct 20. PMID 25329419
- [Background] Canda AE, Sokmen S, Terzi C, Arslan C, Oztop I, Karabulut B, Ozzeybek D, Sarioglu S, Fuzun M. Complications and toxicities after cytoreductive surgery and hyperthermic intraperitoneal chemotherapy. Ann Surg Oncol. 2013 Apr;20(4):1082-7. doi: 10.1245/s10434-012-2853-x. Epub 2013 Mar 2. PMID 23456387
- [Background] Newton AD, Bartlett EK, Karakousis GC. Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy: a review of factors contributing to morbidity and mortality. J Gastrointest Oncol. 2016 Feb;7(1):99-111. doi: 10.3978/j.issn.2078-6891.2015.100. PMID 26941988
- [Background] Hemker HC, Giesen P, AlDieri R, Regnault V, de Smed E, Wagenvoord R, Lecompte T, Beguin S. The calibrated automated thrombogram (CAT): a universal routine test for hyper- and hypocoagulability. Pathophysiol Haemost Thromb. 2002 Sep-Dec;32(5-6):249-53. doi: 10.1159/000073575. PMID 13679651
- [Background] Roest M, van Holten TC, Fleurke GJ, Remijn JA. Platelet Activation Test in Unprocessed Blood (Pac-t-UB) to Monitor Platelet Concentrates and Whole Blood of Thrombocytopenic Patients. Transfus Med Hemother. 2013 Apr;40(2):117-25. doi: 10.1159/000350688. Epub 2013 Mar 28. PMID 23652405
- [Background] Ninivaggi M, Feijge MA, Baaten CC, Kuiper GJ, Marcus MA, Ten Cate H, Lance MD, Heemskerk JW, van der Meijden PE. Additive roles of platelets and fibrinogen in whole-blood fibrin clot formation upon dilution as assessed by thromboelastometry. Thromb Haemost. 2014 Mar 3;111(3):447-57. doi: 10.1160/TH13-06-0493. Epub 2013 Nov 21. PMID 24258426
- [Background] Etulain J, Lapponi MJ, Patrucchi SJ, Romaniuk MA, Benzadon R, Klement GL, Negrotto S, Schattner M. Hyperthermia inhibits platelet hemostatic functions and selectively regulates the release of alpha-granule proteins. J Thromb Haemost. 2011 Aug;9(8):1562-71. doi: 10.1111/j.1538-7836.2011.04394.x. PMID 21649851
- [Background] Cardenas JC, Rahbar E, Pommerening MJ, Baer LA, Matijevic N, Cotton BA, Holcomb JB, Wade CE. Measuring thrombin generation as a tool for predicting hemostatic potential and transfusion requirements following trauma. J Trauma Acute Care Surg. 2014 Dec;77(6):839-45. doi: 10.1097/TA.0000000000000348. PMID 25099452
- [Background] Kuiper GJ, Henskens YM. Rapid and Correct Prediction of Thrombocytopenia and Hypofibrinogenemia with Rotational Thromboelastometry in Cardiac Surgery Reconsidered. J Cardiothorac Vasc Anesth. 2016 Dec;30(6):e55-e56. doi: 10.1053/j.jvca.2016.04.009. Epub 2016 Apr 12. No abstract available. PMID 27498262
- [Background] Perez-Ruixo C, Valenzuela B, Peris JE, Bretcha-Boix P, Escudero-Ortiz V, Farre-Alegre J, Perez-Ruixo JJ. Platelet Dynamics in Peritoneal Carcinomatosis Patients Treated with Cytoreductive Surgery and Hyperthermic Intraperitoneal Oxaliplatin. AAPS J. 2016 Jan;18(1):239-50. doi: 10.1208/s12248-015-9839-0. Epub 2015 Nov 17. PMID 26577587
- [Background] Votanopoulos K, Ihemelandu C, Shen P, Stewart J, Russell G, Levine EA. A comparison of hematologic toxicity profiles after heated intraperitoneal chemotherapy with oxaliplatin and mitomycin C. J Surg Res. 2013 Jan;179(1):e133-9. doi: 10.1016/j.jss.2012.01.015. Epub 2012 Mar 10. PMID 22480844
- [Background] McGovern KF, Lascola KM, Smith SA, Clark-Price SC, McMichael M, Wilkins PA. Assessment of acute moderate hyperglycemia on traditional and thromboelastometry coagulation parameters in healthy adult horses. J Vet Emerg Crit Care (San Antonio). 2012 Oct;22(5):550-7. doi: 10.1111/j.1476-4431.2012.00792.x. Epub 2012 Aug 29. PMID 22931303
- [Background] Gielen CL, Grimbergen J, Klautz RJ, Koopman J, Quax PH. Fibrinogen reduction and coagulation in cardiac surgery: an investigational study. Blood Coagul Fibrinolysis. 2015 Sep;26(6):613-20. doi: 10.1097/MBC.0000000000000307. PMID 26083991
- See also: Hyperthermic intraperitoneal chemotherapy — http://www.cancercenter.com/treatments/hipec/
- Available data/document: Study Protocol — https://drive.google.com/open?id=0B0qo2hDQpXhncWZFZkNfZXhZMjVuUGcxc0IzZll5TEtjaXdn
- Available data/document: Advice Ethical Committee: eudract/B-nr B37120154199 — https://drive.google.com/open?id=0B0qo2hDQpXhnU3AzRHY0d1NtVmlsSmx1cFhKOGtKLTVscno0